CLINICAL TRIAL: NCT04826367
Title: Relaxation Training By Tele-Rehabilitation Program In Patients With Breast Cancer Receiving Chemotherapy During COVID-19.
Brief Title: Relaxation Training by Tele-Rehabilitation in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Umut Bahçacı, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tele-Relax
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Relaxation Therapy; Tele-Rehabilitation; Chemotherapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consists randomly allocated exercise and control groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (EG) (Experimental): The participants in the EG will perform relaxation exercises in groups of up to 8 people, 3 days a week for 6 weeks via WhatsApp (© 2020 WhatsApp, Inc.) or Zoom (© 2012-2020 Zoom Video Communications, Inc.) applications. Relaxation exercises will be performed with the "Progressive Relaxation Exercises (PRE)" technique defined by Jacobson et al.[11] Tele-rehabilitation sessions will last approximately 40 minutes of each, accompanied by a physiotherapist who has 8 years of experience in the field of oncological rehabilitation.
  Interventions: Other: Telerehabilitation-based relaxation exercise group (EG)
- Control Group (CG) (No Intervention): Participants in this group will have a brochure with simple exercises (relaxation exercises involving the upper and lower extremities) in sitting and lying positions. They will be advised to be as active as possible at home and to take mild walks at home. Any supervised exercise program will not apply to participants in the CG. If the participants apply any regular exercise program within 6 weeks, the participants in this group will be excluded from the study.

INTERVENTIONS:
Other: Telerehabilitation-based relaxation exercise group (EG) — the participants in this group will perform the relaxation exercises thrice a week, for 6 weeks.
  Arms: Exercise Group (EG)

SUMMARY:
With developing treatment methods, oncological rehabilitation has become an important complementary part of cancer treatment. Due to the COVID-19 pandemic, the use of tele-rehabilitation has gained importance in terms of access to physical therapy in individuals with breast cancer. Considering the home environment and the patient profile, it is thought that relaxation exercises can be used in the most comfortable and safe way for patients to reduce the side effects of chemotherapy and can be used as home exercises whose effectiveness has been reported in the literature. The purpose of our study; to examine the effects of relaxation exercises performed by tele-rehabilitation on functional capacity, fatigue, emotional state, quality of life, cognitive status, sleep quality and kinesiophobia in breast cancer patients receiving chemotherapy. A total of 64 patients, will randomly be allocated to the exercise group (n = 32) and to the control group (n = 32). Participants will be evaluated at first appoinment and after 6 weeks of intervention. 'Brief Pain Questionnaire' for assessment of pain as assessment methods, 'Fatigue Impact Scale' for fatigue assessment, 'Hospital Anxiety-Depression Scale' for emotional state, 'EORTC QLQ-C30 Quality of Life Scale' for quality of life assessment, 'The FACT-Cog questionnaire' for cognitive state assessment, the' Pitsburg Sleep Quality Scale 'for the measurement of sleep quality, and the' Tampa Kinesophobia Scale 'for the assessment of kinesiophobia will be used.

DETAILED DESCRIPTION:
The study is planned as a single center, single-blind (assessment), randomized and home-based tele-rehabilitation intervention. The study will be conducted at Gayrettepe Florence Nightingale Hospital between January 2021 and November 2022. Participants will consist of individuals with breast cancer undergoing a routine taxane chemotherapy program. The participants will randomly be assigned to study (telerehabilitation-based relaxation exercises) and control groups.

Participants who will meet criteria's will be informed by the medical oncologist involved in the study in the medical oncology clinic in hospital and an informed consent form will be provided to the volunteers who want to participate in the study. After approval of the consent form, participants will be randomly divided into two groups. To provide randomization at a 1:1 sharing ratio, 2 blocks will be created with the "block randomization" method, computer-generated numbers will be put in sealed envelopes. The number from the envelope selected by the patients will indicate which block will be. Randomizations will be made by a non-study researcher. The assessor will also be blind to allocations of the groups. Demographic information of the participants will be recorded and pain, fatigue, emotional state, quality of life, cognitive status, sleep quality and kinesiophobia will be evaluated.

In order to calculate the sample size, power analysis (80% power and 5% type 1 error) was performed with the standard deviation and confidence interval data of the "pain" parameter provided from a reference article[9] similar to this study, The target sample size was determined with the aim of recruiting at least 20 participants per group, based on a power of 80% and a confidence interval of 95%, with an effect size of 0,91. With a possible 30% loss of patient to follow-up was added and totally, it was aimed to include 26 patients in each group.

Assessments will be made at baseline and after 6 weeks of intervention. In case of significant results, exercise programs will be provided to the participants who cannot take the relevant exercises in the control group.

Interventions Telerehabilitation-based relaxation exercise group (EG)

The participants in the EG will perform relaxation exercises in groups of up to 8 people, 3 days a week for 6 weeks via WhatsApp (© 2020 WhatsApp, Inc.) or Zoom (© 2012-2020 Zoom Video Communications, Inc.) applications. Relaxation exercises will be performed with the "Progressive Relaxation Exercises (PRE)" technique defined by Jacobson et al.[11] Tele-rehabilitation sessions will last approximately 40 minutes of each, accompanied by a physiotherapist who has 8 years of experience in the field of oncological rehabilitation. The expected relaxations of the hand, elbow, shoulder, hip, knee, ankle, and facial muscles will be executed by PRE performed throughout the course of the session. Each exercise will be conducted as 5 seconds of contraction and 10 seconds of relaxation. Breathing techniques will occasionally be performed between exercises, so that the effectiveness of relaxation will be increased. The work area will be desired to be well ventilated and an environment where individuals are comfortable. Individuals will be asked to take a long sitting position in comfortable seats. Then, the following instructions will be given to the patients in order:

* Punch your hands and contract your forearm
* Punch your hands, push your elbow towards the seat
* Bend your elbows
* Push your shoulders back
* Press your knee down and pull your toes towards you
* Pull your knees towards you and push your feet down
* Tighten your hips
* Push your head back
* Lift your eyebrows
* Make wrinkles on your nose
* Tighten your teeth
* Push your chin down
* Close your eyes and think of good things. Necessary recommendations for the absence of any factors that create stress during exercise will be given. Patients who miss 10% of the therapy sessions will be excluded from the study.

Control Group (CG) Participants in this group will have a brochure with simple exercises (relaxation exercises involving the upper and lower extremities) in sitting and lying positions. They will be advised to be as active as possible at home and to take mild walks at home. Any supervised exercise program will not apply to participants in the CG. If the participants apply any regular exercise program within 6 weeks, the participants in this group will be excluded from the study.

Outcomes The pain evaluation was identified as the primary outcome, while the fatigue, emotional state, quality of life, cognitive status, sleep quality and kinesiophobia were evaluated as secondary outcomes. Each patient was evaluated in the initial session prior to chemotherapy administration. A subsequent six-week intervention session was then conducted, with the same assessments repeated immediately following the intervention's completion.

Pain assessment: "Brief Pain Inventory (BPİ)" will be used for pain assessment. It is a 9-question scale that evaluates the location and severity of pain, especially with the last 24-hour activities. A validity and reliability study has been performed for the short pain inventory, which is commonly used in cancer patients.[12, 13] Scores between 3-4 are defined as mild pain, between 5-7 as moderate, and between 8-10 as severe pain.

Fatigue assessment: It will be measured with the 'Fatigue Impact Scale (FIS)'. This scale, consisting of 40 items, evaluates the effects of fatigue on physical, cognitive, and psychosocial functions. Higher scores indicate greater exposure to fatigue. Validity and reliability study has been conducted.[14] Emotional state assessment: It will be measured by the "Hospital Anxiety and Depression (HAD)" scale. It is a scale consisting of 14 questions and validity and reliability study has been done.[15] 7 of these questions evaluate anxiety, 7 evaluate depression in this Likert type measurement. The cut-off score for the anxiety subscale is 10/11 and for the depression subscale it is 7/8. Accordingly, those above these scores are considered at risk.

Quality of life assessment: European Organization for Research and Treatment of Cancer- Quality of life (EORTC QLQ-C30) questionnaire will be used to measure the quality of life of individuals. The questionnaire has 3 subtitles and 30 questions: general health, functional score, and symptom score. The first 28 of the 30 items in the scale are a four-point Likert type scale and are scored as 1 (not at all) and 4 (very much) points. Questions 29 and 30 are the form of the domain of general well-being. Higher scores indicate better symptom severity for overall health and functional score, and worse for symptom score. The validation and reliability of the questionnaire was conducted.[16] Cognitive state assessment: Functional Assessment of Chronic Illness Therapy-Cognitive Function (FACT-Cog) will be used to evaluate individuals' cognitive function. The questionnaire, consists of 37 items and 4 different subtitles, evaluates perceived cognitive skills, interpretations of other people, perceived cognitive disorders and quality of life. Individuals determine how valid a certain statement is for them in the last 7 days with a 5-point scale that includes scores between 0 (none) and 4 (very much). Higher scores indicate better cognitive functioning. Validity and reliability study of the questionnaire has been done.[17] Sleep quality: will be measured with the Pittsburg Sleep Quality Index (PSQI). This scale, validity and reliability have been studied, consists of a total of 24 questions with 7 components.[18] These components; subjective sleep quality, time to fall asleep, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime dysfunction. If the total score obtained from these components is above 5, it indicates the "poor sleep" quality. For scores of 5 and below, sleep quality is considered 'good'.

Kinesiophobia evaluation: It will be evaluated with the "Tampa Kinesophobia Scale (TKS)". There are 17 questions in this scale, which was developed to measure the fear of motion / re-injury. 4-point Likert scoring (1 = Strongly disagree, 4 = Strongly agree) is used in the scale. The total score is between 17-68. The high score the person gets on the scale indicates that his kinesiophobia is also high. The validity and reliability study has been done.[19]

Statistical Analysis SPSS version 26.0 (Copyright © IBM Corporation and its licencors 1989, 2019) program will be used for statistical evaluation. A descriptive analysis will be performed and the mean, 95% confidence interval and standard deviations (SDs) will be calculated for each group. Initially, Student's t test and Chi-square test will be used to check for differences between groups. Normal distribution of variables will be analyzed by Shapiro-Wilk test. Intervention effects on study variables will be tested using the repeated measure ANCOVA. If a significant interaction occurs in the analysis, paired comparisons will be made with the Bonferroni test to determine whether there is a difference in scores between groups. Also, the effect size will be calculated using Cohen's d values. P<0.05 will be considered significant.

Anticipated Results:

1) Observing positive effects of relaxation exercises with tele-rehabilitation on pain, fatigue, emotional state, quality of life, cognitive status, sleep quality and kinesophobia in individuals with breast cancer who received chemotherapy during Covid-19 period.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance scale ≥90,
* Age between 18-65,
* Taxan class chemotherapy program has been planned,
* Not having regular exercise habits in the last 6 months,
* Patients who gave consent to voluntarily participate in the study.

Exclusion Criteria:

* Having a communication problem
* Standardized mini mental test score ≤23
* Previous chemotherapy treatments
* Having a neurological, rheumatological or orthopedic problem that prevents working,
* Presence of advanced lymphedema (Stage 3-4),
* Recurrence during treatment,
* Failing to use technology for tele-rehabilitation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | 24 hours
  Assesses the severity of pain and its impact on functioning. Consisting of 17 questions, evaluating pain location, severity, and pain status, especially in the last 24 hours. Scores of 3-4 are defined as mild, 5-7 as moderate, 8-10 as severe pain in this scale.
'Fatigue Impact Scale (FIS) | 1 week
  This scale, consisting of 40 items, evaluates the effects of fatigue on physical, cognitive, and psychosocial functions.Each item is rated on a five-step Likert scale, where 0 = no problems to 4 = extreme problems during the previous month. Ratings are summed to a total score, ranging from 0 to 160, and domain scores range from 0 to 40 for physical and cognitive functioning and 0-80 for the psychosocial functioning. Higher scores indicate greater limitations in functioning.
Hospital Anxiety and Depression (HAD)" scale | 1 week
  It is a scale consisting of 14 questions and validity and reliability study has been done.[15] 7 of these questions evaluate anxiety, 7 evaluate depression in this Likert type measurement. The cut-off score for the anxiety subscale is 10/11 and for the depression subscale it is 7/8. Accordingly, those above these scores are considered at risk.
European Organization for Research and Treatment of Cancer- Quality of life (EORTC QLQ-C30) questionnaire | 1 week
  It is used to measure the quality of life of individuals. The questionnaire has 3 subtitles and 30 questions: general health, functional score, and symptom score. The first 28 of the 30 items in the scale are a four-point Likert type scale and are scored as 1 (not at all) and 4 (very much) points. Questions 29 and 30 are the form of the domain of general well-being. Higher scores indicate better symptom severity for overall health and functional score, and worse for symptom score.
Functional Assessment of Chronic Illness Therapy-Cognitive Function (FACT-Cog) | 1 week
  used to evaluate individuals' cognitive function. The questionnaire, consists of 37 items and 4 different subtitles, evaluates perceived cognitive skills, interpretations of other people, perceived cognitive disorders and quality of life. Individuals determine how valid a certain statement is for them in the last 7 days with a 5-point scale that includes scores between 0 (none) and 4 (very much). Higher scores indicate better cognitive functioning.
Pittsburg Sleep Quality Index (PSQI) | 1 month
  consists of a total of 24 questions with 7 components.[18] These components; subjective sleep quality, time to fall asleep, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime dysfunction. If the total score obtained from these components is above 5, it indicates the "poor sleep" quality. For scores of 5 and below, sleep quality is considered 'good'.
Tampa Kinesophobia Scale (TKS) | 1 month
  There are 17 questions in this scale, which was developed to measure the fear of motion / re-injury. 4-point Likert scoring (1 = Strongly disagree, 4 = Strongly agree) is used in the scale. The total score is between 17-68. The high score the person gets on the scale indicates that his kinesiophobia is also high.

CONTACTS AND LOCATIONS:
Overall Officials: Esat Namal, Asst. Prof., Study Chair — Demiroğlu Bilim University
Locations (1):
- Florence Nightingale Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a recent plan to make IPD available

REFERENCES:
- [Background] Brennan D, Tindall L, Theodoros D, Brown J, Campbell M, Christiana D, Smith D, Cason J, Lee A. A blueprint for telerehabilitation guidelines. Int J Telerehabil. 2010 Oct 27;2(2):31-4. doi: 10.5195/ijt.2010.6063. eCollection 2010 Fall. PMID 25945175
- [Background] Cheville AL, Moynihan T, Herrin J, Loprinzi C, Kroenke K. Effect of Collaborative Telerehabilitation on Functional Impairment and Pain Among Patients With Advanced-Stage Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):644-652. doi: 10.1001/jamaoncol.2019.0011. PMID 30946436
- [Background] Mata MD, Marzo MM, Teixidor P, Caceres C, Enseñat A, Boldó M, et al. Randomized controlled trial on the impact of cognitive telerehabilitation on cognition and quality of life in glioma patients. Annals of Physical and Rehabilitation Medicine. 2018;61:e271.
- [Background] Piraux E, Caty G, Reychler G, Forget P, Deswysen Y. Feasibility and Preliminary Effectiveness of a Tele-Prehabilitation Program in Esophagogastric Cancer Patients. J Clin Med. 2020 Jul 9;9(7):2176. doi: 10.3390/jcm9072176. PMID 32660126
- [Background] van der Kolk NM, de Vries NM, Kessels RPC, Joosten H, Zwinderman AH, Post B, Bloem BR. Effectiveness of home-based and remotely supervised aerobic exercise in Parkinson's disease: a double-blind, randomised controlled trial. Lancet Neurol. 2019 Nov;18(11):998-1008. doi: 10.1016/S1474-4422(19)30285-6. Epub 2019 Sep 11. PMID 31521532
- [Background] Mella-Abarca W, Barraza-Sanchez V, Ramirez-Parada K. Telerehabilitation for people with breast cancer through the COVID-19 pandemic in Chile. Ecancermedicalscience. 2020 Aug 5;14:1085. doi: 10.3332/ecancer.2020.1085. eCollection 2020. PMID 32863879
- [Background] Ariza-Garcia A, Lozano-Lozano M, Galiano-Castillo N, Postigo-Martin P, Arroyo-Morales M, Cantarero-Villanueva I. A Web-Based Exercise System (e-CuidateChemo) to Counter the Side Effects of Chemotherapy in Patients With Breast Cancer: Randomized Controlled Trial. J Med Internet Res. 2019 Jul 24;21(7):e14418. doi: 10.2196/14418. PMID 31342907
- [Background] Galiano-Castillo N, Cantarero-Villanueva I, Fernandez-Lao C, Ariza-Garcia A, Diaz-Rodriguez L, Del-Moral-Avila R, Arroyo-Morales M. Telehealth system: A randomized controlled trial evaluating the impact of an internet-based exercise intervention on quality of life, pain, muscle strength, and fatigue in breast cancer survivors. Cancer. 2016 Oct 15;122(20):3166-3174. doi: 10.1002/cncr.30172. Epub 2016 Jun 22. PMID 27332968
- [Background] Jacobson, E. (1938). Progressive muscle relaxation. J Abnorm Psychol, 75(1), 18.
- [Background] Dicle A, Karayurt O, Dirimese E. Validation of the Turkish version of the Brief Pain Inventory in surgery patients. Pain Manag Nurs. 2009 Jun;10(2):107-113.e2. doi: 10.1016/j.pmn.2008.08.002. PMID 19481050
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007
- [Background] Aydemir O. Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. Turk Psikiyatri Derg. 1997;8:187-280.
- [Background] Guzelant A, Goksel T, Ozkok S, Tasbakan S, Aysan T, Bottomley A. The European Organization for Research and Treatment of Cancer QLQ-C30: an examination into the cultural validity and reliability of the Turkish version of the EORTC QLQ-C30. Eur J Cancer Care (Engl). 2004 May;13(2):135-44. doi: 10.1111/j.1365-2354.2003.00435.x. PMID 15115469
- [Background] Atasavun Uysal S, Yildiz Kabak V, Karakas Y, Karabulut E, Erdan Kocamaz D, Keser I, Ozdemir K, Duger T. Investigation of the validity and reliability of the Turkish version of the Functional Assessment of Cancer Therapy-Cognitive Function in cancer patients. Palliat Support Care. 2022 Oct;20(5):694-700. doi: 10.1017/S147895152100136X. PMID 34470680
- [Background] Agargun M. Pittsburgh uyku kalitesi indeksinin gecerligi ve guvenirligi. Turk Psikiyatri Dergisi. 1996;7:107-15.
- [Background] Yilmaz ÖT, Yakut Y, Uygur F, ULUĞ N. Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği. Fizyoterapi Rehabilitasyon. 2011;22:44-9.
- [Background] Scaturro D, Vitagliani F, Mangano MS, Tomasello S, Sconza C, Respizzi S, Vecchio M, Letizia Mauro G. Effect of Telerehabilitation and Outpatient Rehabilitation in Women with Breast Cancer. J Funct Morphol Kinesiol. 2023 Jul 27;8(3):105. doi: 10.3390/jfmk8030105. PMID 37606400